CLINICAL TRIAL: NCT05294523
Title: Priming Dose of Rocuronium and Milliamperage Value for Supramaximal Stimulation of NeuroMuscular Transmission Monitor
Brief Title: Rocuronium and Supramaximal Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Principal Investigator, Wei Chieh Lai, Principal investigator, Taipei Medical University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: N202109050
Record Dates: First submitted 2022-01-31; First posted 2022-03-24 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Neuromuscular Blockade

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rocuronium priming dose 0.06mg/kg (Active Comparator): Add the priming dose of rocuronium 0.06mg/kg after the first supramaximal stimulation data measured
  Interventions: Procedure: Rocuronium priming dose
- Rocuronium priming dose 0.12mg/kg (Active Comparator): Add the priming dose of rocuronium 0.12mg/kg after the first supramaximal stimulation data measured
  Interventions: Procedure: Rocuronium priming dose
- Rocuronium priming dose 0.18mg/kg (Active Comparator): Add the priming dose of rocuronium 0.18mg/kg after the first supramaximal stimulation data measured
  Interventions: Procedure: Rocuronium priming dose

INTERVENTIONS:
Procedure: Rocuronium priming dose — Add the priming dose of rocuronium after the first supramaximal stimulation data measured

SUMMARY:
To shorten induction time, some anesthesiologist gives a priming dose of muscle relaxant before starting Neuromuscular Transmission monitor (NMT). To properly evaluate neuromuscular function during the surgury, baseline supramaximal stimulation of the monitored nerve is mandatory. Not knowing if the priming dose of muscle relaxant affects the supramaximal stimulation current setting, The investigators designed this study to find out.

DETAILED DESCRIPTION:
The NMT monitor module automatically determines the current needed for the supramaximal stimulus, and maintains this current throughout the procedure.

The supramaximal current is the current above which there is no increase in the evoked muscle response. At this stimulus current, all motor units are firing in response to nerve stimulation. According to previous studies, the current was significantly increased in the presence of edema and peripheral neuropathy. In this study, the route of administration, dosage, dosage regimen, and treatment period are basically the same as the investigators anesthesia department's routine procedure for general anesthesia. The difference will be the time the investigators set between the priming dose to final dose of rocuronium is 2 minutes. The investigators use 2 minutes as the peak effect of rocuronium is 105±36S.

To properly evaluate neuromuscular blockade during the surgery, baseline supramaximal stimulation of the monitored nerve is mandatory. Not knowing if the priming dose of muscle relaxant affects the supramaximal stimulation current setting, the investigators designed this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving general anesthesia and use rocuronium for induction

Exclusion Criteria:

* Muscular disease
* Peripheral neuropathy
* Difficult airway or difficult mask ventilation
* Allergy to study related medication
* Pregnant woman
* < 20-year-old or > 65-year-old
* BMI <18.5 or BMI>24.9

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Supramaximal stimulation value | since general anesthesia induction to endotracheal tube intubation, about 10 minutes
  whether the supramaximal stimulation changs after 2 minutes of priming dose of muscle relaxant use

SECONDARY OUTCOMES:
supramaximal stimulation value change by time | since general anesthesia induction to endotracheal tube intubation, about 10 minutes
  whether the supramaximal stimulation changs have a trend
dose of rocuronium | since general anesthesia induction to endotracheal tube intubation, about 10 minutes
  whether the change of supramaximal stimulation change is muscle relaxant dose responsive
Time to intubation | since general anesthesia induction to endotracheal tube intubation, about 10 minutes
  how long does it take from the full dose of muslce relaxant given to TOF count <2
Intubation condition | since general anesthesia induction to endotracheal tube intubation, about 10 minutes
  the intubation condition with priming method used. Evaluate with scoring scale. scale range from 0-3. 0 presented as poor Jaw relaxation, closed vocal cord, and severe cough or bucking when intubation; to 3 represent a condition with good jaw relaxation, open vocal cord, and no repsponse to stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chieh Lai, MD, MPH, Study Chair — Taipei Medical University Hospital
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
de-identified raw data

REFERENCES:
- [Background] Kopman AF, Lawson D. Milliamperage requirements for supramaximal stimulation of the ulnar nerve with surface electrodes. Anesthesiology. 1984 Jul;61(1):83-5. No abstract available. PMID 6742488
- [Background] Naguib M, Brull SJ, Kopman AF, Hunter JM, Fulesdi B, Arkes HR, Elstein A, Todd MM, Johnson KB. Consensus Statement on Perioperative Use of Neuromuscular Monitoring. Anesth Analg. 2018 Jul;127(1):71-80. doi: 10.1213/ANE.0000000000002670. PMID 29200077
- [Background] Armendariz-Buil I, Lobato-Solores F, Aguilera-Celorrio L, Morros-Diaz E, Fraile-Jimenez E, Vera-Bella J. Residual neuromuscular block in type II diabetes mellitus after rocuronium: a prospective observational study. Eur J Anaesthesiol. 2014 Aug;31(8):411-6. doi: 10.1097/01.EJA.0000435022.91954.8d. PMID 24201596
- [Background] Fuchs-Buder T, Claudius C, Skovgaard LT, Eriksson LI, Mirakhur RK, Viby-Mogensen J; 8th International Neuromuscular Meeting. Good clinical research practice in pharmacodynamic studies of neuromuscular blocking agents II: the Stockholm revision. Acta Anaesthesiol Scand. 2007 Aug;51(7):789-808. doi: 10.1111/j.1399-6576.2007.01352.x. PMID 17635389
- See also: Diabetes Mellitus and Neuromuscular Blockade: Review — https://www.iomcworld.com/open-access/diabetes-mellitus-and-neuromuscular-blockade-review-2155-6156-1000678.pdf